CLINICAL TRIAL: NCT03203746
Title: Gingival Crevicular Fluid Levels of Protein Carbonyl Oxidative Stress Biomarker Following the Use of Locally Delivered Lycopene Antioxidants in Patients With Chronic Periodontitis - Randomized Clinical Trial
Brief Title: Gingival Crevicular Fluid Levels of Protein Carbonyl Following the Use of Lycopene in Chronic Periodontitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Maie Sami tawfik (Other)
Responsible Party: Sponsor-Investigator, Maie Sami tawfik, Principal investigator, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Maie Sami
Record Dates: First submitted 2017-06-24; First posted 2017-06-29 (Actual); Last update posted 2017-06-29 (Actual); Status verified 2017-06

CONDITIONS: Chronic Periodontitis
Keywords: Lycopene; Chronic periodontitis; Protein carbonyl
MeSH Terms: conditions — Chronic Periodontitis | interventions — Lycopene

STUDY DESIGN:
Intervention Model Description: Total subjects selected were allocated into three study groups, Group I (Test group), Group II (Positive control group) and Group III (Negative control group). Group I: Included 8 patients with severe chronic periodontitis managed by Scaling and root planing (SRP) and local delivery of lycopene loaded in solid lipid microparticles. Group II: Included 8 patients with severe chronic periodontitis managed by Scaling and root planing (SRP) only. Group III: Included 8 patients with clinically healthy periodontium.
Masking Description: No masking
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group I: Lycopene + SRP (Experimental): Lycopene, 0.1 ml injected once in the periodontal pocket after scaling and root planing
  Interventions: Drug: Lycopene + SRP
- Group II: SRP only (Active Comparator): Scaling and root planing only without lycopene
  Interventions: Procedure: SRP only
- Group III: healthy subjects (No Intervention): No intervention

INTERVENTIONS:
Drug: Lycopene + SRP
  Arms: Group I: Lycopene + SRP
Procedure: SRP only
  Arms: Group II: SRP only

SUMMARY:
Effect of Locally Delivered Antioxidants as An Adjunct to Non-surgical Periodontal Therapy on GCF Level of Oxidative Stress Marker; Protein Carbonyl

DETAILED DESCRIPTION:
The study was designed as a randomized controlled clinical trial. Total subjects selected were allocated into three study groups, Group I (Test group), Group II (Positive control group) and Group III (Negative control group). Group I: Included 8 patients with severe chronic periodontitis managed by Scaling and root planing and local delivery of lycopene loaded in solid lipid microparticles. Group II: Included 8 patients with severe chronic periodontitis managed by Scaling and root planing only. Group III: Included 8 patients with clinically healthy periodontium.

Protein carbonyl biomarker level and clinical parameters were assisted to evaluate the effect of lycopene as an adjunct to scaling and root planing.

ELIGIBILITY:
Inclusion Criteria:

* All subjects were free from any systemic diseases.
* Subjects for group I and II were suffering from severe chronic periodontitis (Armitage et al., 1999).
* Group III included subjects with clinically healthy periodontium.
* All subjects were between 35-60 years old.
* Both genders were included.
* Subjects were able to return for follow up visits.
* Subjects agreed to sign a written consent after the nature of the study was explained.

Exclusion Criteria:

* History of scaling and root planing or periodontal surgery < 6 months prior to initiation of the study.
* History of administration of antimicrobial drugs or over the counter antioxidants like Vit C, Vit B, β-carotene < 6 months prior to the baseline examination.
* Subjects who reported any side effects or drug allergies from antioxidants.
* Subjects with mobile teeth, abscesses and defected restorations related to the affected sites.
* Subjects with para-functional habits.
* Pregnant and lactating females.
* Smokers, alcoholic and drug abusers.
* Prisoner.
* Mentally retarded patients.

Ages: 35 Years to 52 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2015-09-28 (Actual); Primary Completion 2016-11-10 (Actual); Study Completion 2016-12-14 (Actual)

PRIMARY OUTCOMES:
GCF level of protein carbonyl | 1 month
  to assess GCF level of protein carbonyl following local delivery of sustained release form of lycopene as an adjunct to scaling and root planning (SRP) in management of severe chronic periodontitis patients.

SECONDARY OUTCOMES:
Plaque index | 6 months
  To assess changes in plaque index following local delivery of stained release form of lycopene.
Modified gingival index | 6 months
  to assess changes in the gingival index following local delivery of sustained release form of lycopene.
Probing depth | 6 months
  To assess probing depth following local delivery of stained release form of lycopene.
Clinical attachment loss | 6 minths
  To assess clinical attachment loss following local delivery of sustained release form of lycopene.
Radiographic changes | 6 months
  to assess radiographic changes in the infrabony defects following local delivery of sustained release form of lycopene.
Drug release | 1 month
  to assess rate of lycopene release using high performance liquid chromatography technique (HPLC).

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Y Gamal, PhD, Study Director — AinShams university

IPD SHARING:
Plan to Share IPD: No